CLINICAL TRIAL: NCT02381873
Title: Exploratory Study of Determinants of Early Functional Outcome Following Reconstructive Knee Surgery
Brief Title: Determinants of Early Functional Outcome After Reconstructive Surgery
Status: Completed | Type: Observational
Sponsor: Queen Margaret University (Other)
Responsible Party: Principal Investigator, Maria Peer, PhD Research Student, Queen Margaret University
Other Study IDs: 14/NE/1216
Record Dates: First submitted 2015-02-28; First posted 2015-03-06 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Osteoarthritis
Keywords: Arthroplasty; Replacement; Knee; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood serum samples
Oversight: Data Monitoring Committee: No

SUMMARY:
This exploratory study will quantify and describe patient-reported and objective measures of sensorimotor, neuromuscular, psychophysiological and genotypical performance capabilities and levels of habitual physical activity prior to and around the time of surgery.

DETAILED DESCRIPTION:
Despite the positive outcomes of total knee arthroplasty (TKA) surgery on symptoms such as pain, perceived function and health-related quality of life (QoL) current research highlights the persistent deleterious effects of retained aberrant neuromuscular alterations on physical function, which may also directly impact falls risk. Importantly, observed increases in neuromuscular deficits that occur prior to surgery track through into the post-operative stage with functional limitations that are sustained and which can persist at least one year after surgery. Clearly, it is crucial to strive to identify modifiable factors that might successfully ameliorate this pathophysiological process prior to surgery, reduce post surgical impairments and which also accelerate recovery.

Among other determinants that might contribute towards understanding of optimal functional recovery following reconstructive knee surgery is the influence of genes. The evaluation of specific genotypes and subsequent protein expression might provide further insight into the extent of genetic influence. For example, it is not yet known whether patients with specific genotypes experience an accelerated recovery. Currently, there is a paucity of research on the influence of gene-environment interactions on an individual's response to physical conditioning.

The proposed research will be an exploratory study, involving four repeated-measures assessments from 10 weeks prior to surgery to 12 weeks after surgery. This study offers a novel evaluation of the overall patterning of changes and will quantify and describe patient-reported and objective measures of sensorimotor, neuromuscular, psychophysiological performance capabilities, genotypes and levels of habitual physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Males and females over the age of 18, diagnosed with severe osteoarthritis and awaiting primary TKA.

Exclusion Criteria:

* Individuals electing primary knee arthroplasty surgery due to a knee joint disease other than osteoarthritis
* Rheumatic disorder
* Other orthopaedic conditions affecting lower body function
* Neurological disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females over the age of 18, diagnosed with severe osteoarthritis and awaiting primary total knee arthroplasty (TKA).
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Score (KOOS) | from 10 weeks prior to surgery to 12 weeks after surgery
  Self reported questionnaire which evaluates pain, other symptoms, function in activity of daily living, function in sport and recreation (Sport/Rec), and knee related QoL.
Oxford knee score (OKS) | from 10 weeks prior to surgery to 12 weeks after surgery
  Self reported questionnaire which evaluates pain and function.
Postural stability as assesed by force plate | from 10 weeks prior to surgery to 12 weeks after surgery
  Postural stability will be assessed using a stable force plate.

SECONDARY OUTCOMES:
Neuromuscular performance capability | from 10 weeks prior to surgery to 12 weeks after surgery
  Dynamometer and electromyography measurements will be used to evaluate neuromuscular performance capability.
Sensorimotor performance capability | from 10 weeks prior to surgery to 12 weeks after surgery
  Dynamometer and electromyography measurements will be used to evaluate sensorimotor performance capability.
International Physical Activity Questionnaire (IPAQ). | from 10 weeks prior to surgery to 12 weeks after surgery
  Self-reported physical activity will be monitored using IPAQ.
Knee circumference | from 10 weeks prior to surgery to 12 weeks after surgery
DNA genotypes and subsequent protein expression | on the day of surgery and 12 weeks following operation
Psychophysiological response | from 10 weeks prior to surgery to 12 weeks after surgery
  Self reported. Psychophysiological response will be assessed using Category-Ratio Scale (CR-10); performance profile; short form (SF)-36.

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Peer, Principal Investigator — Queen Margaret University
Locations (1):
- Robert Jones & Agnes Hunt Orthopaedic Hospital NHS Foundation Trust, Oswestry, Shropshire, United Kingdom